CLINICAL TRIAL: NCT02077036
Title: Narcolepsy - New Potential Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Lars Hyllienmark, Associate professor, consultant in neurology and clinical neurophysiology, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: nervus11
Record Dates: First submitted 2014-02-11; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

ARMS (2):
- Active medical device (Experimental)
  Interventions: Device: Kinetic Oscillation Stimulation Device
- Inactive medical device (Placebo Comparator)
  Interventions: Device: Kinetic Oscillation Stimulation Device in placebo mode

INTERVENTIONS:
Device: Kinetic Oscillation Stimulation Device
  Arms: Active medical device
Device: Kinetic Oscillation Stimulation Device in placebo mode
  Arms: Inactive medical device

SUMMARY:
The overall aim of the study is to investigate the effect of a new, non-pharmacological method that may alleviate the symptoms of narcolepsy and thereby lead to a reduction in the use of medications with potentially serious side effects in patients with this disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosed with narcolepsy (diagnose code G47.4)
* 16 - 60 years of age
* MSLT has shown hypersomnia (sleeping latency < 8 min) & 1 episode REM
* HLA-type associated with increased occurrence of narcolepsy

Exclusion Criteria:

* Reduced cognitive function
* Other relevant organ disease (that could affect the study results or put the patient at risk)
* Ongoing bacterial infection in the nose
* Comorbidity that can increase the risk of bleeding
* Has received treatment with an implantable stimulator or other implantable product in the head and / or in the neck
* Known pronounced septal deviation
* Known allergy to polyvinylchloride or medicinal liquid paraffin
* Women not using adequate contraceptives
* Participated in a clinical investigational drug trial within the previous 30 days

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in scale Epworth Sleep Scale (ESS) | 15-21 days
  Change in ESS scale between baseline before treatment and at 15-21 days after treatment.

SECONDARY OUTCOMES:
Change in multiple sleep latency test (MSLT) | 14 days
  Change in MSLT (mean sleep latency, number of sleep onset rapid eye movement (SOREM), and mean SOREM latency) between registration at baseline and 14 days after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden